CLINICAL TRIAL: NCT02493894
Title: By Reza Abbasi and Isfahan University of Medical Sciences
Brief Title: The Effect of Bowel Preparation on Perioperative Bleeding
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Isfahan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Abbasi, Dr. Abbasi, Isfahan University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Abbasi1
Record Dates: First submitted 2015-06-18; First posted 2015-07-10 (Estimated); Last update posted 2015-07-10 (Estimated); Status verified 2015-07

CONDITIONS: Surgery
Keywords: Bowel preparation; perioperative bleeding; lumbar fusion
MeSH Terms: interventions — polyethylene glycol 3350; salicylhydroxamic acid; Cefazolin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PEG & Cefazolin (Experimental): patients firstly get liquid diet for 24 hours. After that they get PEG solution (80gr/1Litr) each 8 hours for 24 hours. After 48 hours, cefazolin 1gram, every 6hours for 2 days
  Interventions: Drug: PEG; Drug: Cefazolin
- placebo & cefazolin (Sham Comparator): placebo for PEG and cefazolin 1gram, every 6hours for 2 days
  Interventions: Drug: placebo; Drug: Cefazolin

INTERVENTIONS:
Drug: PEG — PEG solution (80gr/1Litr) each 8 hours for 24 hours
  Other Names: PEG solution
  Arms: PEG & Cefazolin
Drug: placebo — placebo each 8 hours for 24 hours
  Other Names: sham
  Arms: placebo & cefazolin
Drug: Cefazolin — cefazolin 1gram, every 6hours for 2 days
  Other Names: Kefzol

SUMMARY:
Now a days, due to the change in lifestyle, the extended lifespan and the increase in the rate of the road accidents, the need for surgical operation of spinal instrumentation has been increased. And these surgeries are the most crucial part of neurological surgery wards. The everyday improvements in the quality of equipment used and advancements in surgical methods lead to best performance of these procedures and finally the higher quality of patients' lives. The procedures of Laminectomy and pedicular screw instrumentation lead to pain relief and better performance and developments in the quality of patients' lives.

In addition to the above mentioned improvements, you must consider the fact that these activities are still accompanied by complications during and after surgical operation.

Nerve root injury, Thecal sac tearing, injury to the spinal cord and the inappropriate sagittal balance are the most significant side effects during spinal surgery.

One of the most important complications during and after these surgeries is perioperative bleeding that causes problems both for the patients and the surgeon.

DETAILED DESCRIPTION:
The individuals evaluated in this study were those who have been admitted and undergone spiral surgery (Fusion and Instrumentation) with pedicular screw because of spinal column instability and canal stenosis.

This study has been started and performed since Feb.2013 to June 2015 at the neurosurgery ward of Al.zahra hospital of Isfahan.

The candidates chosen for the study were those who undergone the surgery procedure due to degenerative change of Lumbar spinal canal.

The necessity of operation for each patient is diagnosed based on clinical finding, Imaging data and guidelines according to neurosurgery reference sources.(Richards Winn,Youmans Neurological Survey, Sixth Edition, Vol 3,Ch.303) During this prospective study, patients are randomly divided into two groups of Case and Control. The individuals attended these two groups are matched regarding age, sex and general medical condition. The age ranges in this study are 33 to 82 years old.

Other than general surgery consent taken from both groups, patients in Case group are informed about the procedure of the program and probable side effects.

Primarily, patients' weight, height, BMI, and Hemoglobin are recorded. In Case group, patients firstly get liquid diet for 24 hours. After that they get PEG solution (80gr/1Litr) each 8 hours for 24 hours. After 48 hours, bowel is mechanically prepared for the procedure. Cefazolin 1 gram every 6hours for 2 days was taken in both groups.

In both Case and Control groups, the time of surgery and the volume of bleeding (in CC) are precisely recorded by surgery and anesthesiology team. The need for blood transfusion during surgery is based on preoperation hemoglobin and the volume of bleeding during surgery and is calculated according to anesthesiology and surgical standards using the following formula:

( )/Hb ×0.6 BW kg×10022 Immediately at the end of surgery, the exact rate of bleeding during operation ( in CC), the length of operation and the length of the operation and the estimated transfusion rate are recorded.

Also, after surgery the volume of bleeding in homovac drain in time intervals of 24 to 48-hour are recorded.

Also the patients' levels of Hb in 24 to 48-hour intervals are calculated. After improving general medical conditions of the patients and their walking abilities, they are ambulated and finally are discharged from hospital.

ELIGIBILITY:
Inclusion Criteria:

* Patients who suffer from lumbar spine degenerative disease and need spine fusion surgery.

Exclusion Criteria:

* History of Trauma,
* History of Malignancy,
* previous spinal surgery,
* History of coagulation disorder,
* active infectious disease,
* gastrointestinal problems,
* severe movement disorders.

Ages: 33 Years to 82 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2014-07; Primary Completion 2015-05 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
The volume of bleeding was measured in milliliter | up to 3 days

CONTACTS AND LOCATIONS:
Overall Officials: Reza Abbasi, MD, Principal Investigator — Alzahra University Hospital
Locations (1):
- Alzahra Hospital, Isfahan, Isfahan, Iran

REFERENCES:
- [Result] Zhang F, Wang K, Li FN, Huang X, Li Q, Chen Z, Tang YB, Shen HX, Song QX. Effectiveness of tranexamic acid in reducing blood loss in spinal surgery: a meta-analysis. BMC Musculoskelet Disord. 2014 Dec 22;15:448. doi: 10.1186/1471-2474-15-448. PMID 25532706
- See also: http://www.ncbi.nlm.nih.gov/pmc/articles/PMC4326491/ — http://www.ncbi.nlm.nih.gov/pubmed/25532706